CLINICAL TRIAL: NCT03929523
Title: End-ischemic Hypothermic Oxygenated Perfusion for Extended Criteria Donors in Liver Transplantation - A Multicenter, Randomized Controlled Trial
Brief Title: Hypothermic Oxygenated Perfusion for Extended Criteria Donors in Liver Transplantation (HOPExt)
Acronym: HOPExt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0034; 2019-A00546-51 (Other: ANSM)
Record Dates: First submitted 2019-04-09; First posted 2019-04-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Liver Transplantation
Keywords: Liver Transplantation; Liver machine perfusion; extended criteria donor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOPE group (Experimental): hypothermic oxygenated perfusion
  Interventions: Device: End-ischemic Hypothermic Oxygenated Machine Perfusion (HOPE)
- Control group (Active Comparator): classic static cold storage
  Interventions: Device: classic static cold storage

INTERVENTIONS:
Device: End-ischemic Hypothermic Oxygenated Machine Perfusion (HOPE) — In the experimental group, ECD liver grafts will first undergo a classical static cold (4°C) storage with Institute George Lopez (IGL-1)® solution from graft harvesting until transport to the transplantation center. They will then undergo a hypothermic oxygenated perfusion (HOPE) via the portal vein for a period of 1 to 4 hours (minimum 1 hour) after the "back-table" phase (graft preparation), in parallel with the recipient hepatectomy, using the CE-certified Liver Assist® perfusion pump/device (Organ Assist®, the Netherlands) with Machine Perfusion Solution (Belzer-MPS, CE-certified).
  Arms: HOPE group
Device: classic static cold storage — The control group will consist of a classic static cold (4°C) storage with Institute George Lopez (IGL-1)® solution from graft harvesting until liver transplantation, which is the gold standard procedure in liver transplantation
  Arms: Control group

SUMMARY:
Given the scarce donor supply, an increasing number of so-called marginal or extended criteria donor (ECD) organs have been used for liver transplantation. These ECD liver grafts are, however, known to be associated with a higher rate of early allograft dysfunction (EAD) and primary non-function because of a greater vulnerability to ischemia-reperfusion injury. The end-ischemic Hypothermic Oxygenated Machine Perfusion (HOPE) technique may improve outcomes of liver transplantation with ECD grafts by decreasing reperfusion injury.

The study aim is to assess the efficacy of HOPE used before transplantation of ECD liver grafts from brain-dead donors in reducing postoperative EAD within the first 7 postoperative days (POD) compared to simple cold static storage.

The study is comparative open-label, multicenter, national, prospective, randomized, in two parallel groups, using the gold standard procedure as control.

DETAILED DESCRIPTION:
This multicentric randomized controlled trial concerns adult patients undergoing whole liver transplantation in any of the 8 participating centers in France, who will receive an ECD liver graft from a brain-dead donor.

After providing written informed consent prior to the performance of any study specific procedure, the recruited patients will be randomized either in the experimental group (HOPE group) or in the control group.

In the HOPE group, ECD liver grafts will undergo a hypothermic oxygenated perfusion (HOPE) via the portal vein for a period of 1 to 4 hours (minimum 1 hour) after the "back-table" phase (graft preparation), in parallel with the recipient hepatectomy, using the CE-certified Liver Assist® perfusion pump/device (Organ Assist®, the Netherlands) with Machine Perfusion Solution (Belzer-MPS, CE-certified).

The control group will consist of a classic static cold (4°C) storage with Institute George Lopez (IGL-1)® solution from graft harvesting until liver transplantation, which is the gold standard procedure in liver transplantation.

The primary endpoint will be early allograft dysfunction (EAD) according to Olthoff's criteria, which will be compared with the Model of Early Allograft Function score (MEAF score) and the Liver Graft Assessment Following Transplantation risk factor (L-GrAFT).

According to the primary endpoint, a sample size of 133 patients per randomized group (266 in total) is needed. The duration of the inclusion period is expected to be 36 months with a 1-year follow-up for each patient.

The potential impacts of the study are expected on 3 levels: (1) for the patient, decreased postoperative morbidity and mortality of liver transplantation with ECD donors; (2) for the French liver transplantation community, familiarization with liver machine perfusion, and (3) economically, decreased costs of liver transplantation (health economic analysis included in the study).

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to the performance of any study specific procedure
* Affiliated to the French social security system
* Recipient age ≥ 18 years
* Patients undergoing primary liver transplantation.
* Candidate for a first elective liver transplantation, whatever the indication, with a liver graft harvested from a brain-dead ECD defined by the presence of at least one of the following criteria:

  * Donor age > 65 years
  * Intensive care unit stay > 7 days
  * BMI > 30
  * Proven macro-steatosis biopsy ≥ 30%
  * Natremia > 155 mmol/L at any time
  * AST > 150 IU/mL at any time
  * ALT > 170 IU/mL at any time.

Exclusion Criteria:

* Fulminant hepatic failure
* Retransplantation
* Split liver transplantation
* Living donor liver transplantation
* Grafts donated after cardiac arrest (DCD grafts)
* Domino transplantation
* Combined liver transplant
* Unexpected medical contraindication to liver transplantation
* Patient participating in other interventional research, excluding routine care research (old regulation) and category 2 research not interfering with primary endpoint analysis
* Patient under legal protection
* Patient deprived of liberty by a judicial or administrative decision
* Patient refusing to participate in the study
* Pregnant or lactating women
* Inability to understand information concerning the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Early allograft dysfunction (EAD) according to Olthoff criteria. | During the first postoperative week
  EAD is defined by the presence of at least one of the following criteria:
  * Bilirubin level > 10 mg/dL (i.e. 171 µmol/L) on POD 7
  * International Normalized Ratio (INR) > 1.6 on POD 7
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels > 2000 IU/L within the first 7 PODs Additionally EAD will be also assessed by the MEAF score and the L-GrAFT risk factor.

SECONDARY OUTCOMES:
Model of Early Allograft Function score (MEAF score). | During the first 3 postoperative days.
  The MEAF score includes bilirubin, ALT max and INR max at postperative day 3. Range 0 (better outcome) to 10 (worse outcome)
Liver Graft Assessment Following Transplantation risk factor (L-GrAFT) | During the first 10 postoperative days.
  L-GrAFT includes aspartate aminotransferase (AST), INR, total bilirubin and platelets every day until postoperative day 10. Range -6 (better outcome) to +6 (worse outcome)
Untargeted liver graft metabolic profiling | Day of liver transplantation (Day 0)
  Untargeted liver graft metabolic profiling (by High-Resolution Nuclear Magnetic Resonance - 1H HR-Nuclear Magnetic Resonance (NMR) Spectrometer) on liver graft biopsies on the back-table before and after liver machine perfusion.
Occurrence of post-reperfusion syndrome | Day of liver transplantation (Day 0)
  Defined as a 50% decrease in median arterial pressure during the 5 minutes following the graft revascularization
90-day morbidity and mortality | During the first 90 days after surgery.
  Severe postoperative complications (Dindo-Clavien ≥3) / death
Length of intermediate care unit stay (days) | From randomization until intermediate care unit discharge, estimated up to 7 days
  Duration of intermediate care unit stay
Length of hospital stay (days) | From randomization until hospital discharge, estimated up to 21 days
  Duration of hospital stay
Liver contrast-enhanced MRI including a Magnetic Resonance CholangioPancreatography (MRCP) | Within 1 year after liver transplantation
  Assessment of intra- and extrahepatic biliary complications (except for patients who underwent a re-transplanted during the study).
3-month and one-year patient and graft survivals | within one year after liver transplantation
  Actuarial graft and patient's survival rates
Hospital costs (Euros) of liver transplantation | At one year after liver transplantation
  Hospital costs of liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Mickael LESURTEL, Principal Investigator — APHP Beaujon
Locations (8):
- France (8):
  - Department of HPB surgery and liver transplantation Beaujon University Hospital, Clichy
  - CHU Grenoble Alpes - Department of HPB surgery and liver transplantation, Grenoble
  - Department of HPB surgery and liver transplantation Claude Huriez University Hospital, Lille
  - Hospices Civils de Lyon, Lyon
  - APHP - Pitié Salpétrière, Paris
  - Department of HPB surgery and liver transplantation Pontchaillou University Hospital, Rennes
  - Hôpital Hautepierre - Department of HPB surgery and liver transplantation, Strasbourg
  - Department of HPB surgery and liver transplantation Paul Brousse University Hospital, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pradat P, Pantel S, Maynard M, Lalande L, Thevenon S, Adam R, Allard MA, Robin F, Rayar M, Boleslawski E, Scatton O, Chirica M, Faitot F, Bachellier P, Soubrane O, Mohkam K, Mabrut JY, Lesurtel M. End-ischemic hypothermic oxygenated perfusion for extended criteria donors in liver transplantation: a multicenter, randomized controlled trial-HOPExt. Trials. 2023 Jun 6;24(1):379. doi: 10.1186/s13063-023-07402-0. PMID 37280696
- [Result] Lesurtel M, Mohkam K, Allard MA, Adam R, Robin F, Rayar M, Boudjema K, Chebaro A, Boleslawski E, Savier E, Scatton O, Girard E, Chirica M, Dokmak S, Soubrane O, Faitot F, Bachellier P, Hervieu V, Guerre P, Atfeh J, Pantel S, Thevenon S, Maynard M, Pradat P, Mabrut JY. A French multicenter randomized controlled trial of hypothermic oxygenated perfusion in extended criteria donor liver transplantation. Am J Transplant. 2025 Oct 17:S1600-6135(25)03053-9. doi: 10.1016/j.ajt.2025.10.006. Online ahead of print. PMID 41110608